CLINICAL TRIAL: NCT06913842
Title: Adrenal Myelolipomas Case Series Laparoscopic Management
Brief Title: Adrenal Myelolipomas Case Series
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Huber Díaz Fuentes, Urologist, Instituto Mexicano del Seguro Social
Other Study IDs: 98235522
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Adrenal Myelolipoma
Keywords: Adrenal, Incidentaloma, Myelolipoma, Laparoscopy.
MeSH Terms: conditions — Myelolipoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Six cases (72 years old female patient, 63 years old male patient, 57 years old female patient, 61 years old female, 72 years old female and 56 years old female) of clinically and radiologically suspected cases of symptomatic adrenal myelolipoma are discussed here. All cases described, presented with flank pain radiating which was suspected as adrenal mass by Computed Tomography (CT) evaluation. All six cases were histopathologically confirmed as adrenal myelolipoma and managed by laparoscopic surgical excision.

DETAILED DESCRIPTION:
The management in all cases was by laparoscopic adrenalectomy with transperitoneal approach. Several retrospective and comparative studies addressed the advantage of minimally invasive adrenalectomy specifically consistent in less postoperative pain, improved patients' satisfaction, shorter hospital stay and recovery time when compared to open adrenalectomy.

The laparoscopic transabdominal lateral adrenalectomy is currently the most widely used approach.

All our cases were managed by this technique. In our cases initial peritoneal access is achieved 2cm inferior to the right/left costal margin in the midclavicular line, a pressure of 15mmHg is used for CO2 insufflation. Optical access 10-12mm trocar for the endoscope is placed in the pararectal line 5cm above the umbilicus. Under direct vision, the second 10- 12 mm trocar is placed medially to the first one. The third trocar (5mm) is inserted 3 cm above the anterior superior iliac spine in the anterior axillary line. The fourth trocar (5mm) is inserted at the subcostal angle. The key factor for an adequate exposure is an effective dissection of the Toldt fascia. Vascular structures are ligated with Hem-O-Lock and subsequent dissection of the adrenal gland with ultrasonic energy. The adrenal is extracted through a Gibson-type incision, a Penrose drain was left in all cases with its removal upon discharge of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adrenal myelolipoma

Exclusion Criteria:

* Patients without CT scan with myelolipoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 6 Patients who underwent laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months
  Mortality in surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Mexican Social Security Institute: Regional General Hospital No. 1, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Anyone who ask via E-mail.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Samimagham H, Kazemi Jahromi M. Bilateral Adrenal Myelolipoma, A Case Presentation and Brief Literature Review. Iran J Kidney Dis. 2020 Jan;14(1):62-64. PMID 32156843